CLINICAL TRIAL: NCT03321786
Title: Legionella Pneumonia's Effect on Olfactory Function
Brief Title: Legionnaires' Effect on Smell
Status: Completed | Type: Observational
Sponsor: University of Pennsylvania (Other)
Responsible Party: Principal Investigator, Richard Doty, Director, Smell and Taste Center, Professor of Psychology in Otorhinolaryngology: Head and Neck Surgery, University of Pennsylvania
Other Study IDs: 827730
Record Dates: First submitted 2017-10-23; First posted 2017-10-26 (Actual); Last update posted 2024-07-24 (Actual); Status verified 2024-07

CONDITIONS: Legionnaires' Disease
MeSH Terms: conditions — Legionnaires' Disease

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Legionnaires' Disease Volunteers: Volunteers who have been diagnosed/survivors of Legionnaire's Disease
  Interventions: Other: The University of Pennsylvania Smell Identification Test (UPSIT)
- Healthy Volunteers: Volunteers who are healthy.
  Interventions: Other: The University of Pennsylvania Smell Identification Test (UPSIT)

INTERVENTIONS:
Other: The University of Pennsylvania Smell Identification Test (UPSIT) — This standardized test, the most widely used olfactory test in the world, is derived from basic psychological test measurement theory and focuses on the comparative ability of subjects to identify odorants at the suprathreshold level. The UPSIT consists of four envelope-sized booklets, each containing ten "scratch and sniff" odorants embedded in 10- 50-µm polymer microcapsules positioned on brown strips at the bottom of the pages of the booklets.

SUMMARY:
The goal of this study is to determine whether survivors of Legionnaires' disease suffer smell loss. A quantitative olfactory test will be performed by the participants. Such testing will require approximately 20-30 minutes of the participant's time. The participants will take the University of Pennsylvania Smell Identification Test (UPSIT), a scratch-and-sniff test to assess their ability to identify odors in a forced- choice format. Volunteers will also complete a questionnaire asking personal history, demographic questions, and medical history.

ELIGIBILITY:
Inclusion Criteria:

* Persons of generally good health, as obtained from a screening questionnaire who are 18 years of age and older
* Both men and women of all ethnic backgrounds will be accepted.

Exclusion Criteria:

* Age less than 18
* Pregnant Women
* Persons who mental competence is limited, such as those with dementia

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: The subjects to be tested in this study represent two different populations. The first is a group of who have survived Legionnaires' disease. The second group will be healthy men and women over the age of 18 years.
Sampling Method: Non-Probability Sample
Enrollment: 10 (Actual)
Dates: Start 2017-09-06 (Actual); Primary Completion 2024-06-15 (Actual); Study Completion 2024-06-15 (Actual)

PRIMARY OUTCOMES:
Score on the University of Pennsylvania Smell Identification Test | 20-30 Minutes
  The number of correct odor identification responses out of 40 from the standardized University of Pennsylvania Smell Identification Test.
  The total number of correct responses will then be compared to standard norms of correct responses based on demographic information such as age and sex. Comparing the scores to the standard norms collected will indicate whether a volunteer is normosmic, hyposmic, or anosmic.

SECONDARY OUTCOMES:
Questionnaire Responses | 20-30 Minutes
  These are various demographic and medical history questions regarding exposure to Legionella Pneumonia and current experiences post diagnosis and treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Richard L Doty, PhD, Principal Investigator — University of Pennsylvania
Locations (1):
- University of Pennsylvania, Philadelphia, Pennsylvania, United States